CLINICAL TRIAL: NCT05572827
Title: The Efficiency of Breathing Exercises Performed on COVID-19 Patients After Intensive Care
Brief Title: The Efficiency of Breathing Exercises
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ataturk University (Other)
Responsible Party: Principal Investigator, Bahar Ciftci, Principal Investigator, Ataturk University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: Atatürk U
Record Dates: First submitted 2022-09-15; First posted 2022-10-10 (Actual); Last update posted 2023-01-09 (Actual); Status verified 2023-01

CONDITIONS: Breathing Exercises
MeSH Terms: interventions — Breathing Exercises

STUDY DESIGN:
Who Masked: Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental (Experimental): Breathing exercises will be taught to COVID-19 patients after intensive care.
  Interventions: Behavioral: Breathing exercises
- Control (No Intervention): Breathing exercises will not be taught to COVID-19 patients after intensive care.

INTERVENTIONS:
Behavioral: Breathing exercises — Breathing exercises for COVID-19 patients after intensive care increase their quality of life.
  Arms: Experimental

SUMMARY:
The purpose of this study is to evaluate the effectiveness of teaching breathing exercises to COVID-19 patients after intensive care.The research is a randomized controlled and pretest-posttest applied design. The population of the research will consist of patients who have been previously admitted to the intensive care unit of the hospital where the research will be conducted and who meet the research criteria.The data of the study are "Patient Information Form" and "Data Registration Form", "Care dependency scale", "Health Screening short form-36", "Saint George Respiratory Questionnaire (SGRQ), "Respiratory Function Test", "Respiratory Exercises Information Booklet" and "Breathing Exercises Information Booklet".

DETAILED DESCRIPTION:
Aim of research The purpose of this study is to evaluate the effectiveness of teaching breathing exercises to COVID-19 patients after intensive care.

Type of research The research is a randomized controlled and pretest-posttest applied design. Research Population and Sample Selection The population of the research will consist of patients who have been previously admitted to the intensive care unit of the hospital where the research will be conducted and who meet the research criteria. In order to determine the sample size, a priori power analysis was performed and it was determined that at least 35 patients were required for each of the intervention and control groups in order for the power of the study to exceed 80% at the 95% confidence interval, 0.05 significance level and medium effect size. Considering that there may be data loss due to various reasons, 80 patients are planned to be included in the sample of the study.

Data collection tools and features The data of the study are "Patient Information Form" and "Data Registration Form", "Care dependency scale", "Health Screening short form-36", "Saint George Respiratory Questionnaire (SGRQ), "Respiratory Function Test", "Respiratory Exercises Information Booklet" and "Breathing Exercises Information Booklet".

1. Data Registration Form. It is the form in which the blood pressure, pulse, respiration, body temperature, oxygen saturation values taken twice a day, before and after exercise, are recorded.
2. Patient Identification Form. Patients have name-surname, age, gender, height, weight, BMI, educational status, occupation, marital status, clinical data (history, family history, medications used, use of assistive devices, smoking history, respiratory system evaluation) and exercise habits.
3. Care dependency scale. In the study, this scale was used to determine the care dependency of the patients.

   The lowest score obtained from the scale is 17 and the highest score is 85. A high scale score indicates that the individual is independent in meeting their care needs, while a low scale score indicates that the individual is dependent on meeting their care needs.
4. Baseline dyspnea scale Mahler et al. It was developed by 1984. The validity and reliability of the Basal Dyspnea Scale in our country have been made by different researchers, and the scale evaluates dyspnea due to activity; It measures in three different areas: functional status (level of performing activities of daily living), effort capacity (difficult efforts to perform activities) and work capacity.
5. Health Screening short form-36 Short Form-36 (Short Form-36 Health Survey - SF-36) will be used to assess overall health-related quality of life. SF-36 is a self-rating scale. Subscales evaluate health on a scale of 0-100, with 0 indicating poor health and 100 indicating good health.
6. Saint George Respiratory Questionnaire (SGRQ) The Saint George Respiratory Questionnaire (SGRQ) will be used to assess the disease-specific quality of life. The SGRQ is a questionnaire in which patients self-answer questions. The questionnaire, which consists of three categories, questions the effects of symptoms, activity and illness on daily life. It is considered to be more standardized than other health-related quality of life questionnaires. It is mostly used in COPD, asthma and bronchiectasis. It has an evaluation scale between 0-100 points in the questionnaire consisting of a total of 76 questions. Zero indicates best health and 100 indicates worst health.
7. Pulmonary Function Test Pulmonary function tests are an objective method used in the diagnosis and follow-up of the disease. Pulmonary function tests were performed in a sitting position with a computer compatible spirometer

Research Intervention Materials Breathing Exercises Information Booklet; Respiratory Exercises Information Booklet created by the researchers in line with the literature review; It includes information about the disease and its treatment, treatment methods of the disease, lifestyle changes that are effective in respiratory management, and the importance of compliance with treatment.

Breathing Exercises Video CDs; The content will be created by the researchers in line with the literature review. Videos; It includes information about the disease and its treatment, treatment methods of the disease, lifestyle changes that are effective in respiratory management, and the importance of compliance with treatment. The content of the training booklet and the training videos will be the same.

Data Collection All patients in the intervention and control groups who meet the inclusion criteria will be verbally informed about the purpose of the study and the method of application. "Informed Consent Form" will be filled in for the patients who agree to participate in the study. Then, pre-test forms ("Patient Identification Form", "Care dependency scale", "Health Screening short form-36", "Saint George Respiratory Questionnaire (SGRQ)) will be filled in by face-to-face interview method for all patients in the intervention and control groups.

Randomization in the study will be determined randomly by using a computer program (researcher randomizer), provided that the number of individuals in the intervention and control groups is equal regardless of the characteristics of the participants such as age and gender.

Enterprise Group; The vital signs of the patients in the intervention group, for which the necessary forms are filled, will be taken and the "Data Registration Form" will be filled. Afterwards, patients will have Pulmonary Function Tests and the results will be filled in the "Respiratory Function Test Report". Afterwards, breathing exercises will be taught in line with the "Respiratory Exercises Information Booklet" and "Respiratory Exercises Information Booklet". As long as the patients stay in the hospital, it will be checked whether they do their exercises. When the patients are completely discharged, they will be called by phone and reminded to do their exercises three times a day.

In this way, patients in the intervention group will be followed remotely by tele-nursing for 8 weeks. At the end of the 8th week, the patients will be called to the hospital and the recorded data will be received from the patients. Then, as a posttest, the patients will have Pulmonary Function Tests and the results will be filled in the "Respiratory Function Test Report". Likewise, as posttest ("Care dependency scale", "Health Screening short form-36", "Saint George Respiratory Questionnaire (SGRQ)) forms will be filled again.

control group; No intervention will be made in the control group. For the final test, the results will be filled into the "Respiratory Function Test Report" after 8 weeks. Likewise, as posttest ("Care dependency scale", "Health Screening short form-36", "Saint George Respiratory Questionnaire (SGRQ)) forms will be filled again.

Evaluation of data The data will be evaluated in the SPSS (Statistical Package for Social Sciences for Windows, Version 22.0) package program.

Research Ethics Ethical permission was obtained from the Ethics Committee of Atatürk University Faculty of Medicine for the study to be carried out. Institutional permission was obtained from the hospital where the research would be conducted. In addition, informed consent will be obtained from the participants who agree to participate in the study. The research will be in accordance with the Declaration of Helsinki.

ELIGIBILITY:
Inclusion Criteria:

1. Being a patient who was treated in the intensive care unit and referred to the clinic due to Covid-19 PCR positivity
2. Ability to do exercises appropriately
3. Absence of any communication or medically defined mental problems
4. Being able to understand and speak Turkish
5. Not having any disease that may be risky for the study (uncontrolled diabetes, malignant hypertension, thyrotoxicosis, orthopedic defect, muscle and joint disease)
6. Volunteering to participate in the study

Exclusion Criteria:

1. Not being treated in the intensive care unit due to Covid-19 PCR positivity
2. Having any communication or medically defined mental problems
3. Inability to properly perform exercises prepared for study
4. Those with an uncontrollable additional disease (diabetes, thyrotoxicosis, malignant hypertension)
5. Those who cannot understand and speak Turkish
6. Refusal to participate in the study

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2022-10-01 (Actual); Study Completion 2022-12-01 (Actual)

PRIMARY OUTCOMES:
Data Registration Form. | 3 months
  It is the form in which the systolic blood pressure, diastolic blood pressure, pulse, respiration, body temperature, oxygen saturation values taken twice a day, before and after exercise, are recorded.
Patient Identification Form. | 3 months
  Patients have name-surname, age, gender, height, weight, educational status, occupation, marital status, clinical data (history, family history, medications used, use of assistive devices, smoking history, respiratory system evaluation) and exercise habits.
Baseline dyspnea scale | 3 months
  Mahler et al. It was developed by 1984. The validity and reliability of the Basal Dyspnea Scale in our country have been made by different researchers, and the scale evaluates dyspnea due to activity; It measures in three different areas: functional status (level of performing activities of daily living), effort capacity (difficult efforts to perform activities) and work capacity.
Health Screening short form-36 Short Form-36 | 3 months
  (Short Form-36 Health Survey - SF-36) will be used to assess overall health-related quality of life. SF-36 is a self-rating scale. Subscales evaluate health on a scale of 0-100, with 0 indicating poor health and 100 indicating good health.
Saint George Respiratory Questionnaire (SGRQ) | 3 months
  The Saint George Respiratory Questionnaire (SGRQ) will be used to assess the disease-specific quality of life. The SGRQ is a questionnaire in which patients self-answer questions. The questionnaire, which consists of three categories, questions the effects of symptoms, activity and illness on daily life. It is considered to be more standardized than other health-related quality of life questionnaires. It is mostly used in COPD, asthma and bronchiectasis. It has an evaluation scale between 0-100 points in the questionnaire consisting of a total of 76 questions. Zero indicates best health and 100 indicates worst health.
Pulmonary Function Test | 3 months
  Pulmonary function tests are an objective method used in the diagnosis and follow-up of the disease. In pulmonary function tests, the percentages of forced expiratory volume in the first second (FEV1), forced vital capacity (FVC), the ratio of forced expiratory volume in the first second to forced vital capacity (FEV1/FVC), peak flow rate (PEF), values to the expected value will be recorded.
Care dependency scale. | 3 months
  In the study, this scale was used to determine the care dependency of the patients.
  The lowest score obtained from the scale is 17 and the highest score is 85. A high scale score indicates that the individual is independent in meeting their care needs, while a low scale score indicates that the individual is dependent on meeting their care needs.

CONTACTS AND LOCATIONS:
Overall Officials: Bahar Çiftçi, Study Director — Ataturk University
Locations (1):
- Atatürk University Faculty of Nursing, Erzurum, Turkey (Türkiye)